CLINICAL TRIAL: NCT05726487
Title: ACTION (physicAl aCtiviTy In minOrity womeN With Asthma) Intervention: Efficacy to Implementation
Brief Title: Physical Activity Intervention for Black Women With Asthma
Acronym: ACTION E2I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of Illinois at Chicago (Other); University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB22-0911
Record Dates: First submitted 2023-01-11; First posted 2023-02-14 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-04

CONDITIONS: Asthma
Keywords: Black women; Asthma Control Questionnaire; Physical Activity
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTION Intervention (Experimental): Orientation (week 0): 1 group session Induction phase (weeks 1-12): 8 weekly then 2 bi-weekly goal setting via text with health coach + 2 group sessions (week 5, 9) Adoptive phase (weeks 13-24): 2 monthly goal setting with remote health coach + 3 group sessions (week 13, 17, 21) Maintenance phase (weeks 25-48): 1 group session Outcome assessment (12-, 24-, and 48-weeks)
  Interventions: Behavioral: ACTION Intervention
- Education Control (Other): Orientation (week 0): 1 individual asthma education session Education texts: weekly (weeks 1-8), then bi-weekly (week 9-12), then monthly (weeks 13-24) Outcome assessments (12-, 24-, 48-weeks)
  Interventions: Other: Education Control

INTERVENTIONS:
Behavioral: ACTION Intervention — Participants in the ACTION Intervention arm of the study will have group sessions, physical activity self-monitoring, text-based support for goal setting. Following this intervention participants will be followed for an additional 24-weeks to assess for the maintenance of intervention effects on asthma health outcomes.
  Arms: ACTION Intervention
Other: Education Control — Participants in the Education Control arm of the study will receive and individual asthma education session and text messages related to asthma education. Following this intervention participants will be followed for an additional 24-weeks to assess for the maintenance of intervention effects on asthma health outcomes.
  Arms: Education Control

SUMMARY:
Physical inactivity is associated with poor asthma control and quality of life, and greater health care utilization. Rates of physical inactivity, asthma, and asthma mortality among Black women are higher than those of their White counterparts. Our formative work identified barriers to PA among Black women with asthma including a lack of social support, self-efficacy, unsafe neighborhood and fear related to experiences with life-threatening asthma exacerbations. Given the unique barriers to PA and high rates of physical inactivity that are associated with poor asthma outcomes in Black women, there is an urgent need to optimize PA interventions for this population. The proposed study uses our theory-driven intervention (ACTION: A lifestyle physiCal acTivity Intervention for minOrity womeN with asthma) to deliver a 24-week lifestyle physical activity intervention designed for and by urban Black women with asthma. Participants will be recruited through two urban health care systems that care for a diverse urban Black populations. Participants will be randomized to one of two groups: 1) ACTION intervention (group sessions, physical activity self-monitoring and text-based support for goal-setting), or 2) education control (an individual asthma education session and text messages related to asthma education). Participants will be followed for an additional 24-weeks after the intervention to assess for the maintenance of intervention effects on asthma health outcomes. We are proposing an efficacy study that focuses on asthma outcomes (Aim 1A/B), explores behavioral mechanisms of the intervention (Aim 2) and assesses factors that influence its reach and implementation potential (Aim 3). This trial will provide the first ever evidence of the efficacy of a lifestyle physical activity intervention among urban Black women with asthma, a population that is understudied yet plagued by low levels of PA and poor health outcomes. Our study has high potential to advance clinical treatment of asthma, and further the mechanistic understanding of physical activity interventions in minority populations living in low-resourced urban environments.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as female and Black or African-American
* Age >/= 18
* Physician-diagnosed persistent asthma that is sub-optimally controlled based on Asthma Control Test (ACT < 20) OR history in the past year of an asthma exacerbation (a need for systemic corticosteroids or hospital admission or emergency treatment for worsening asthma)
* Willing to enroll and provide written-informed consent
* Willing to be randomly assigned to treatment or control group
* Low- active: engages in less than 150 minutes per week of moderate-to- vigorous physical activity
* Has a smartphone and texts every day or almost everyday

Exclusion Criteria:

* Plans to relocate outside of the Chicagoland area during the study period
* Unable to ambulate without the use of a wheelchair or scooter
* Diagnosis of COPD (emphysema or chronic bronchitis) suggested by patient report of doctor diagnosis or smoking history (≥ 20 pack years)
* Current tobacco smoker
* A contraindication to exercise as indicated by the Physical Activity Readiness Questionnaire unless written permission by a health care provider
* Significant medical (e.g., unstable heart disease, uncontrolled high blood pressure, active cancer treatment in past 1 year, end-stage organ failure) or psychiatric (e.g., active bipolar disorder, psychosis) comorbidities
* Participation in another physical activity or asthma research program
* Asthma exacerbation, defined by an urgent care visit for asthma in the last 4 weeks, or need for acute course of systemic corticosteroids for asthma in the last 4 weeks
* Family/household member of another study participant or staff member
* Inability to speak, read or understand English
* Investigator discretion for safety or protocol adherence reasons
* Unable or unwilling to provide complete accelerometry data at the baseline assessment after two opportunities to wear the monitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Questionnaire | 24-weeks
  Validated questionnaire

SECONDARY OUTCOMES:
Asthma Control Questionnaire | 48-weeks
  Validated questionnaire
Mini-asthma quality of life questionnaire | 24- and 48-weeks
  Validated questionnaire
Asthma exacerbations | 24- and 48-weeks
  Self-reported measure
Healthcare Utilization (ED, urgent care, and hospitalizations) | 24- and 48-weeks
  Self-reported measure
Self-efficacy for walking scale | 24- and 48-weeks
  Survey
Social support for exercise | 24- and 48-weeks
  Survey
Self-regulation | 24- and 48-weeks
  Measured by exercise self-regulation questionnaire (SRQ-E) and step goals achieved
Light Physical Activity | 24-weeks
  Physical activity measure. Measured by Actigraph GT3XP-BTLE waist-based Accelerometer.
Moderate Physical Activity | 24-weeks
  Physical activity measure. Measured by Actigraph GT3XP-BTLE waist-based Accelerometer.
Moderate-Vigorous Physical Activity | 24-weeks
  Physical activity measure. Measured by Actigraph GT3XP-BTLE waist-based Accelerometer.
Vigorous Physical Activity | 24-weeks
  Physical activity measure. Measured by Actigraph GT3XP-BTLE waist-based Accelerometer.
Daily Steps | 24-weeks
  Physical activity measure. Measured by Actigraph GT3XP-BTLE waist-based Accelerometer
PWMAQ | 24-weeks
  Physical activity measure. Validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sharmilee Nyenhuis, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Illinois Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Avallone KM, McLeish AC. Asthma and aerobic exercise: a review of the empirical literature. J Asthma. 2013 Mar;50(2):109-16. doi: 10.3109/02770903.2012.759963. Epub 2013 Jan 31. PMID 23252987
- [Background] Garcia-Aymerich J, Varraso R, Anto JM, Camargo CA Jr. Prospective study of physical activity and risk of asthma exacerbations in older women. Am J Respir Crit Care Med. 2009 Jun 1;179(11):999-1003. doi: 10.1164/rccm.200812-1929OC. Epub 2009 Feb 26. PMID 19246716
- [Background] Hansen ESH, Pitzner-Fabricius A, Toennesen LL, Rasmusen HK, Hostrup M, Hellsten Y, Backer V, Henriksen M. Effect of aerobic exercise training on asthma in adults: a systematic review and meta-analysis. Eur Respir J. 2020 Jul 30;56(1):2000146. doi: 10.1183/13993003.00146-2020. Print 2020 Jul. PMID 32350100
- [Background] Carson KV, Chandratilleke MG, Picot J, Brinn MP, Esterman AJ, Smith BJ. Physical training for asthma. Cochrane Database Syst Rev. 2013 Sep 30;2013(9):CD001116. doi: 10.1002/14651858.CD001116.pub4. PMID 24085631
- [Background] Kuder MM, Clark M, Cooley C, Prieto-Centurion V, Danley A, Riley I, Siddiqi A, Weller K, Kitsiou S, Nyenhuis SM. A Systematic Review of the Effect of Physical Activity on Asthma Outcomes. J Allergy Clin Immunol Pract. 2021 Sep;9(9):3407-3421.e8. doi: 10.1016/j.jaip.2021.04.048. Epub 2021 May 6. PMID 33964510
- [Background] Akinbami LJ, Moorman JE, Bailey C, Zahran HS, King M, Johnson CA, Liu X. Trends in asthma prevalence, health care use, and mortality in the United States, 2001-2010. NCHS Data Brief. 2012 May;(94):1-8. PMID 22617340
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Nyenhuis SM, Shah N, Ma J, Marquez DX, Wilbur J, Cattamanchi A, Sharp LK. Identifying Barriers to Physical Activity Among African American Women with Asthma. Cogent Med. 2019;6(1):1582399. Epub 2019 Feb 27. PMID 31754624
- [Background] Joseph RP, Ainsworth BE, Keller C, Dodgson JE. Barriers to Physical Activity Among African American Women: An Integrative Review of the Literature. Women Health. 2015;55(6):679-99. doi: 10.1080/03630242.2015.1039184. Epub 2015 Apr 24. PMID 25909603
- [Background] Nyenhuis SM, Balbim GM, Ma J, Marquez DX, Wilbur J, Sharp LK, Kitsiou S. A Walking Intervention Supplemented With Mobile Health Technology in Low-Active Urban African American Women With Asthma: Proof-of-Concept Study. JMIR Form Res. 2020 Mar 11;4(3):e13900. doi: 10.2196/13900. PMID 32159520
- [Background] Nyenhuis SM, Dixon AE, Ma J. Impact of Lifestyle Interventions Targeting Healthy Diet, Physical Activity, and Weight Loss on Asthma in Adults: What Is the Evidence? J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):751-763. doi: 10.1016/j.jaip.2017.10.026. Epub 2017 Dec 6. PMID 29221919
- [Background] Luten KA, Dijkstra A, Reijneveld SA, de Winter AF. Moderators of physical activity and healthy eating in an integrated community-based intervention for older adults. Eur J Public Health. 2016 Aug;26(4):645-50. doi: 10.1093/eurpub/ckw051. Epub 2016 Apr 19. PMID 27095795
- [Background] Clark NM, Valerio MA, Gong ZM. Self-regulation and women with asthma. Curr Opin Allergy Clin Immunol. 2008 Jun;8(3):222-7. doi: 10.1097/ACI.0b013e3282fe9d05. PMID 18560296
- [Background] Piercy KL, Troiano RP, Ballard RM, Carlson SA, Fulton JE, Galuska DA, George SM, Olson RD. The Physical Activity Guidelines for Americans. JAMA. 2018 Nov 20;320(19):2020-2028. doi: 10.1001/jama.2018.14854. PMID 30418471
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Background] National Center for Health Statistics Health, D.o.H.a.H. Services, Editor. 2007: Hyattsville, MD.
- [Background] Ried-Larsen M, Brond JC, Brage S, Hansen BH, Grydeland M, Andersen LB, Moller NC. Mechanical and free living comparisons of four generations of the Actigraph activity monitor. Int J Behav Nutr Phys Act. 2012 Sep 12;9:113. doi: 10.1186/1479-5868-9-113. PMID 22971175
- [Background] Choi L, Liu Z, Matthews CE, Buchowski MS. Validation of accelerometer wear and nonwear time classification algorithm. Med Sci Sports Exerc. 2011 Feb;43(2):357-64. doi: 10.1249/MSS.0b013e3181ed61a3. PMID 20581716
- [Background] Sasaki JE, John D, Freedson PS. Validation and comparison of ActiGraph activity monitors. J Sci Med Sport. 2011 Sep;14(5):411-6. doi: 10.1016/j.jsams.2011.04.003. Epub 2011 May 25. PMID 21616714
- [Background] Prince SA, Cardilli L, Reed JL, Saunders TJ, Kite C, Douillette K, Fournier K, Buckley JP. A comparison of self-reported and device measured sedentary behaviour in adults: a systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2020 Mar 4;17(1):31. doi: 10.1186/s12966-020-00938-3. PMID 32131845
- [Background] Kriska AM, Knowler WC, LaPorte RE, Drash AL, Wing RR, Blair SN, Bennett PH, Kuller LH. Development of questionnaire to examine relationship of physical activity and diabetes in Pima Indians. Diabetes Care. 1990 Apr;13(4):401-11. doi: 10.2337/diacare.13.4.401. PMID 2318100
- [Background] Pereira MA, FitzerGerald SJ, Gregg EW, Joswiak ML, Ryan WJ, Suminski RR, Utter AC, Zmuda JM. A collection of Physical Activity Questionnaires for health-related research. Med Sci Sports Exerc. 1997 Jun;29(6 Suppl):S1-205. No abstract available. PMID 9243481
- [Background] Pettee Gabriel K, McClain JJ, Lee CD, Swan PD, Alvar BA, Mitros MR, Ainsworth BE. Evaluation of physical activity measures used in middle-aged women. Med Sci Sports Exerc. 2009 Jul;41(7):1403-12. doi: 10.1249/MSS.0b013e31819b2482. PMID 19516161
- [Background] Pettee Gabriel K, McClain JJ, Schmid KK, Storti KL, Ainsworth BE. Reliability and convergent validity of the past-week Modifiable Activity Questionnaire. Public Health Nutr. 2011 Mar;14(3):435-42. doi: 10.1017/S1368980010002612. Epub 2010 Sep 15. PMID 20843404
- [Background] Cerin E, Saelens BE, Sallis JF, Frank LD. Neighborhood Environment Walkability Scale: validity and development of a short form. Med Sci Sports Exerc. 2006 Sep;38(9):1682-91. doi: 10.1249/01.mss.0000227639.83607.4d. PMID 16960531
- [Background] Bauman AE, Reis RS, Sallis JF, Wells JC, Loos RJ, Martin BW; Lancet Physical Activity Series Working Group. Correlates of physical activity: why are some people physically active and others not? Lancet. 2012 Jul 21;380(9838):258-71. doi: 10.1016/S0140-6736(12)60735-1. PMID 22818938
- [Background] Harley AE, Rice J, Walker R, Strath SJ, Quintiliani LM, Bennett GG. Physically active, low-income African American women: an exploration of activity maintenance in the context of sociodemographic factors associated with inactivity. Women Health. 2014;54(4):354-72. doi: 10.1080/03630242.2014.896440. PMID 24617833
- [Background] Cooley C, Park Y, Ajilore O, Leow A, Nyenhuis SM. Impact of interventions targeting anxiety and depression in adults with asthma. J Asthma. 2022 Feb;59(2):273-287. doi: 10.1080/02770903.2020.1847927. Epub 2020 Nov 28. PMID 33176512
- [Background] Dixon, A.E.N., S.N. , Obesity and Asthma, in UptoDate, H. Hollingsworth, Editor. 2020, UptoDate: Waltham, MA.
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A; American College of Sports Medicine; American Heart Association. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1081-93. doi: 10.1161/CIRCULATIONAHA.107.185649. Epub 2007 Aug 1. PMID 17671237
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Background] Nici L, Donner C, Wouters E, Zuwallack R, Ambrosino N, Bourbeau J, Carone M, Celli B, Engelen M, Fahy B, Garvey C, Goldstein R, Gosselink R, Lareau S, MacIntyre N, Maltais F, Morgan M, O'Donnell D, Prefault C, Reardon J, Rochester C, Schols A, Singh S, Troosters T; ATS/ERS Pulmonary Rehabilitation Writing Committee. American Thoracic Society/European Respiratory Society statement on pulmonary rehabilitation. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1390-413. doi: 10.1164/rccm.200508-1211ST. No abstract available. PMID 16760357
- [Background] Durstine JL, M.G., Painter P, and Roberts S., ed. ACSM's Exercise Management for Persons with Chronic Diseases and Disabilities. 2009, Human Kinetics: Champaign, IL. 146-148.
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] S, F., User's Manual for ATLAS.ti 5.0. 2004, Scientific Software Development: Berlin.
- [Background] Kvale, S., Inter Views: An introduction to qualitative research interviewing. 1996, Thousand Oaks, CA: Sage.
- [Background] Conrad, P., The experience of illiness: Recent and new directions, in The experience and management of chronic illness, C.P. Roth JA, Editor. 1987, JAI Press: Greenwich, CT.
- [Background] Pacheco JA, Avila PC, Thompson JA, Law M, Quraishi JA, Greiman AK, Just EM, Kho A. A highly specific algorithm for identifying asthma cases and controls for genome-wide association studies. AMIA Annu Symp Proc. 2009 Nov 14;2009:497-501. PMID 20351906
- [Background] Afshar M, Press VG, Robison RG, Kho AN, Bandi S, Biswas A, Avila PC, Kumar HVM, Yu B, Naureckas ET, Nyenhuis SM, Codispoti CD. A computable phenotype for asthma case identification in adult and pediatric patients: External validation in the Chicago Area Patient-Outcomes Research Network (CAPriCORN). J Asthma. 2018 Sep;55(9):1035-1042. doi: 10.1080/02770903.2017.1389952. Epub 2017 Nov 10. PMID 29027824
- [Derived] Davis E, Townsend E, Cavalier A, Chen YF, Edwards-Hart D, Kitsiou S, Kowalczyk W, Mansur I, Okpara E, Powell K, Press VG, Ramirez T, Salvo D, Sharp LK, Wright B, Nyenhuis SM. Physical Activity Intervention for Urban Black Women With Asthma: Protocol for a Randomized Controlled Efficacy Study. JMIR Res Protoc. 2024 Feb 7;13:e55700. doi: 10.2196/55700. PMID 38324365